CLINICAL TRIAL: NCT04820309
Title: An Open-label Study to Assess the Long-term Safety, Tolerability, and Efficacy of KarXT in De Novo Subjects With DSM-5 Schizophrenia
Brief Title: An Open-label Study to Assess the Long-term Safety, Tolerability, and Efficacy of KarXT in Adult Patients With Schizophrenia (EMERGENT-5)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0007; CN012-0007 (Other: Bristol-Myers Squibb Protocol ID); KAR-011 (Other: Karuna Pharmaceuticals Protocol ID)
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KarXT (Experimental)
  Interventions: Drug: Xanomeline and Trospium Chloride Capsules

INTERVENTIONS:
Drug: Xanomeline and Trospium Chloride Capsules — Oral xanomeline 50 mg/trospium 20 mg BID on days 1-2 followed by xanomeline 100 mg/trospium 20 mg BID on days 3-7. The dose is increased to xanomeline 125 mg/trospium 30 mg BID on days 8-364 unless the subject is experiencing adverse events from the xanomeline 100 mg/ trospium 20 mg dose. Subjects who were increased to xanomeline 125 mg/trospium 30 mg will have the option to return to xanomeline 100 mg/ trospium 20 mg depending on clinical response and tolerability. Re-escalation to 125/30 BID or re-titration in cases in which the subject has been off KarXT for a longer period of time (at least a week) is allowed and will require a discussion between the principal investigator and the medical monitor.
  Other Names: KarXT

SUMMARY:
This is a Phase 3, multicenter, 56-week, outpatient, open-label (OL) study to evaluate the long-term safety, tolerability, and efficacy of KarXT in de novo subjects with Diagnostic and Statistical Manual-Fifth Edition (DSM-5) schizophrenia. In this OL study, all subjects will receive KarXT (a fixed combination of xanomeline 125 mg and trospium chloride 30 mg twice daily [BID]) for up to 52 weeks. The primary objective of the study is to assess the long-term safety and tolerability of KarXT in subjects with a DSM-5 diagnosis of schizophrenia. The secondary objective of this study is to assess the long-term efficacy and characterize the pharmacokinetics of xanomeline and trospium after administration of KarXT.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 to 65 years at screening.
2. Subject is capable of providing informed consent.

   1. A signed informed consent form (ICF) must be provided before any study assessments are performed.
   2. Subject must be fluent in (oral and written) the language of the ICGF to consent.
3. Subject has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the DSM-5 (American Psychiatric Association 2013) criteria and confirmed by Mini International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorder Studies (MINI) version 7.0.2.
4. Subject has not required psychiatric hospitalization, acute crisis intervention, or other increase in level of care due to symptom exacerbation within 8 weeks of screening and is psychiatrically stable in the opinion of the investigator.
5. PANSS total score ≤ 80 at screening and Baseline Visit B (Day 0).
6. Clinical Global Impression - Severity (CGI-S) score of ≤ 4 at screening and Baseline Visit B (Day 0).
7. At the time of screening, or at any time within the 30 days prior to screening, the subject must have received an oral antipsychotic medication daily at a dose and frequency consistent with the drug label.
8. In the opinion of the investigator, it is clinically appropriate for the subject to discontinue current antipsychotic therapy and initiate experimental treatment with KarXT.
9. Subject is willing and able, in the opinion of the investigator, to discontinue all antipsychotic medications prior to baseline visit.
10. Subject has an identified reliable informant willing to be able to address some questions related to certain study visits, if needed. An informant may not be necessary if the subject has been the patient of the investigator for ≥1 year.
11. At Day 0, subject will have been off lithium therapy for at least 2 weeks and must have discontinued all oral antipsychotic medications.
12. Subjects taking a long-acting injectable antipsychotic could not have received a dose of medication for at least 12 weeks (24 weeks for paliperidone palmitate) before Day 0.
13. Body mass index must be ≥ 18 and ≤ 40 kg/m2.
14. Subject resides in a stable living situation and is anticipated to remain in a stable living situation for the duration of study enrollment, in the opinion of the investigator.
15. Women of childbearing potential or men with sexual partners of childbearing potential must be willing and able to use at least 1 highly effective method of contraception during the study and for at least 30 days after the last dose of KarXT. Sperm donation is not allowed for 30 days after the final dose of KarXT.

Exclusion Criteria:

1. Any primary DSM-5 disorder other than schizophrenia within 12 months before screening (confirmed using MINI version 7.0.2 at screening).
2. Subject has a history of moderate to severe alcohol use disorder or a substance (other than nicotine or caffeine) use disorder within the past 12 months or a positive urine drug screen (UDS) for a substance other than cannabis at screening or baseline.
3. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results
4. Subject has human immunodeficiency virus (HIV), cirrhosis, biliary duct abnormalities, hepatobiliary carcinoma, and/or active hepatic viral infections based on either medical history or liver function test results.
5. History or high risk of urinary retention, gastric retention, or narrow-angle glaucoma
6. History of irritable bowel syndrome (with or without constipation) or serious constipation requiring treatment within the last 6 months
7. Risk for suicidal behavior during the study as determined by the investigator's clinical assessment and Columbia-Suicide Severity Rating Scale (C-SSRS).
8. Clinically significant abnormal finding from the physical examination, medical history, ECG, or clinical laboratory results at screening.
9. Subjects cannot currently (within 5 half-lives before Day 0) be receiving monoamine oxidase inhibitors, anticonvulsants, tricyclic antidepressants, centrally active anticholinergics, or any other psychoactive medications other than daily antipsychotic maintenance therapy. As-needed anxiolytics and/or sleep aids are permitted. Selective serotonin reuptake inhibitors and serotonin-norepinephrine reuptake inhibitors taken at stable dose may be permitted.
10. Subject has a history of treatment resistance to schizophrenia medications defined as failure to respond to 2 adequate courses of pharmacotherapy (a minimum of 4 weeks at an adequate dose per the label) within the past 12 months or having received clozapine within the past 3 years
11. Pregnant, lactating, or less than 3 months postpartum.
12. If, in the opinion of the investigator (and/or Sponsor), subject is unsuitable for enrollment in the study or subject has any finding that, in the view of the investigator (and/or Sponsor), may compromise the safety of the subject or affect his/her ability to adhere to the protocol visit schedule or fulfill visit requirements.
13. Subjects has tested positive for coronavirus disease 2019 (COVID-19) within 2 weeks of screening.
14. Subject has extreme concerns relating to global pandemics, such as COVID-19, that preclude study participation.
15. Subject has had psychiatric hospitalization(s) for more than 30 days (cumulative) within the 6 months before screening.
16. Subject has prior exposure to KarXT.
17. Risk of violent or destructive behavior.
18. Current involuntary hospitalization or incarceration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb; Inder Kaul, MD, Study Director — Karuna Therapeutics
Locations (116):
- United States (115):
  - Local Institution - 011-238, Little Rock, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Local Institution - 011-201, Rogers, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Local Institution - 011-240, Anaheim, California
  - Advanced Research Center, Inc., Anaheim, California
  - Clinical Innovations, Inc, Bellflower, California
  - Local Institution - 011-222, Bellflower, California
  - Local Institution - 011-263, Bellflower, California
  - Local Institution - 011-257, Cerritos, California
  - ATP Clinical Research Inc, Costa Mesa, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Local Institution - 011-206, Culver City, California
  - ProScience Research Group, Culver City, California
  - Local Institution - 011-253, Garden Grove, California
  - Local Institution - 011-202, Glendale, California
  - Behavioral Clinical Research, Inc., Glendale, California
  - Omega Clinical Trials, La Habra, California
  - Alliance for Wellness dba Alliance for Research, Long Beach, California
  - Alliance for Wellness, Long Beach, California
  - North County Clinical Research (NCCR), Oceanside, California
  - Excell Research Inc, Oceanside, California
  - Local Institution - 011-229, Oceanside, California
  - Local Institution - 011-242, Orange, California
  - NRC Research Institute, Orange, California
  - CNRI-Los Angeles, LLC, Pico Rivera, California
  - Local Institution - 011-244, Pico Rivera, California
  - CITrials, Riverside, California
  - Local Institution - 011-233, Riverside, California
  - CITrials, Santa Ana, California
  - Local Institution - 011-251, Santa Rosa, California
  - Siyan Clinical Research, Santa Rosa, California
  - Local Institution - 011-246, Sherman Oaks, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Collaborative Neuroscience Research, Torrance, California
  - Local Institution - 011-252, Torrance, California
  - Local Institution - 011-224, Hallandale, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Local Institution - 011-261, Hollywood, Florida
  - Homestead Research Institute, Inc., Homestead, Florida
  - Local Institution - 011-231, Homestead, Florida
  - Local Institution - 011-203, Miami, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - Central Miami Medical Institute, Miami, Florida
  - Local Institution - 011-215, Miami, Florida
  - Local Institution - 011-220, Miami, Florida
  - Phoenix Medical Research, Miami, Florida
  - Innovative Clinical Research, Miami Lakes, Florida
  - Local Institution - 011-234, Miami Lakes, Florida
  - Research Centers of America at Fort Lauderdale Behavioral Health Center, Oakland Park, Florida
  - Health Synergy Clinical Research, Okeechobee, Florida
  - Local Institution - 011-216, Okeechobee, Florida
  - Local Institution - 011-219, Pembroke Pines, Florida
  - Pines Care Research Center, Pembroke Pines, Florida
  - Local Institution - 011-262, West Palm Beach, Florida
  - Neuroscience Research Institute, West Palm Beach, Florida
  - Local Institution - 011-259, Atlanta, Georgia
  - Synexus Clinical Research US, Inc., Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Local Institution - 011-237, Atlanta, Georgia
  - Local Institution - 011-235, Decatur, Georgia
  - Local Institution - 011-204, Chicago, Illinois
  - Uptown Research Institute, Chicago, Illinois
  - Local Institution - 011-223, Wichita, Kansas
  - Ascension Via Christi Research, Wichita, Kansas
  - Local Institution - 011-205, Shreveport, Louisiana
  - Louisiana Clinical Research, Shreveport, Louisiana
  - CBH Health, LLC, Gaithersburg, Maryland
  - Local Institution - 011-211, Gaithersburg, Maryland
  - Local Institution - 011-232, Ann Arbor, Michigan
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Local Institution - 011-226, Flowood, Mississippi
  - Precise Research Centers, Flowood, Mississippi
  - Local Institution - 011-227, Saint Charles, Missouri
  - Midwest Research Group - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - St. Charles Psychiatric Associates/Midwest Research Group, Saint Charles, Missouri
  - Arch Clinical Trials, St Louis, Missouri
  - Local Institution - 011-241, St Louis, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - Local Institution - 011-239, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Local Institution - 011-230, Berlin, New Jersey
  - Hassman Research Institute, Marlton, New Jersey
  - Local Institution - 011-249, Marlton, New Jersey
  - Local Institution - 011-256, New York, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Local Institution - 011-210, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Local Institution - 011-250, Rochester, New York
  - Clinical Trials of America, Hickory, North Carolina
  - Local Institution - 011-218, Dayton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Local Institution - 011-248, North Canton, Ohio
  - Neuro-Behavioral Clinical Research, Inc, North Canton, Ohio
  - Cincy Science, West Chester, Ohio
  - Local Institution - 011-221, West Chester, Ohio
  - SP Research PLLC, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Global Medical Institutes LLC Scranton Medical Institute, Moosic, Pennsylvania
  - Local Institution - 011-207, West Chester, Pennsylvania
  - Psychiatric Consultants, Franklin, Tennessee
  - Community Clinical Research, Austin, Texas
  - Local Institution - 011-243, Austin, Texas
  - BioBehavioral Research of Austin P.C., Austin, Texas
  - BioBehavioral Research of Austin, Austin, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Local Institution - 011-236, DeSoto, Texas
  - Local Institution - 011-258, Fort Worth, Texas
  - Core Clinical Research, Richmond, Texas
  - healthTx, Richmond, Texas
  - Cedar Clinical Research, Draper, Utah
  - Local Institution - 011-209, Bellevue, Washington
  - Northwest Clinical Research Center, Bellevue, Washington
  - Local Institution - 011-260, Everett, Washington
- INSPIRA Clinical Research, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Groups:
- KarXT: All subjects started on a lead-in dose of KarXT 50/20 (50 mg xanomeline/20 mg trospium chloride) BID for the first 2 days (Days 1 and 2), followed by KarXT 100/20 BID for the remainder of Week 1 (Days 3 to 7). Dosing was titrated upwards on Day 8 to KarXT 125/30 BID unless the subject was continuing to experience AEs from the previous dose (KarXT 100/20 BID). All subjects who had their dose increased to KarXT 125/30 BID, depending on tolerability, had the option to return to KarXT 100/20 BID. Re-escalation to 125/30 BID or re-titration in cases in which the subject had been off KarXT for a longer period of time (at least 7 days) were allowed.
Period: Overall Study
Arm/Group | KarXT
Started | 566
Completed | 277
Not Completed | 289
Not completed — Adverse Event | 96
Not completed — ineligible for further treatment according to inclusion/exclusion criteria | 1
Not completed — Consent Withdrawn | 93
Not completed — failure to adhere to protocol | 32
Not completed — alcohol or drug use | 6
Not completed — Lost to Follow-up | 46
Not completed — Death | 2
Not completed — Pregnancy | 1
Not completed — Other reasons | 12

BASELINE CHARACTERISTICS:
Arm/Group | KarXT
Number analyzed (Participants) | 566
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.4 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191
  Male | 375
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 119
  Not Hispanic or Latino | 443
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 389
  White | 164
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as events with an onset date on or after the first dose of KarXT. An Adverse Event is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at baseline, worsens during the study, regardless of the suspected cause of the event using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 566
Participants | 466

2. Secondary Outcome: Number of Participants With Serious Treatment Emergent Adverse Events (STEAEs)
Description: An SAE is any untoward medical occurrence, in the view of either the investigator or sponsor, that results in death; is life-threatening; results in inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity, and/or; is a congenital anomaly/birth defect using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 566
Participants | 41

3. Secondary Outcome: Number of Participants With TEAE Leading to Study Drug Discontinuation
Description: as for outcome 1
Time Frame: From time of consent to end of study (approximately 400 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 566
Participants | 100

4. Secondary Outcome: Change From Baseline in PANSS Total Score at Week 52
Description: The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. The positive symptoms in schizophrenia are the excess or distortion of normal function and the negative symptoms are the diminution or loss of normal functions. PANSS total score is the sum of all 30 items with a minimum score of 30 and a maximum score of 210. Higher scores indicate more severe symptoms.
Time Frame: At baseline and week 52
Population: All treated participants with baseline and week 52 PANSS total scores.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | KarXT
Number analyzed (Participants) | 283
Score on a Scale | -5.5 (11.11)

5. Secondary Outcome: Change From Baseline in PANSS Positive Score at Week 52
Description: PANSS positive score is the sum of all PANSS 7 positive symptom scales with a minimum score of 7 and a maximum score of 49. Higher scores indicate more severe symptoms. Participants are rated from 1 to 7 on each symptom scale. The positive symptoms in schizophrenia are the excess or distortion of normal function such as hallucinations, delusions, grandiosity, and hostility.
Time Frame: At baseline and week 52
Population: All treated participants with baseline and week 52 PANSS positive scores.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | KarXT
Number analyzed (Participants) | 283
Score on a Scale | -1.9 (3.71)

6. Secondary Outcome: Change From Baseline in PANSS Negative Score at Week 52
Description: PANSS negative score is the sum of all PANSS 7 negative symptom scales with a minimum score of 7 and a maximum score of 49. Higher scores indicate more severe symptoms. Participants are rated from 1 to 7 on each symptom scale. The negative symptoms in schizophrenia are the diminution or loss of normal functions.
Time Frame: At baseline and week 52
Population: All treated participants with baseline and week 52 PANSS negative scores.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | KarXT
Number analyzed (Participants) | 283
Score on a Scale | -0.8 (4.42)

7. Secondary Outcome: Change From Baseline in PANSS Marder Factor Negative Score at Week 52
Description: PANSS Marder factor score is a subscale of the PANSS; the sum of 5 negative scales and 2 general scales (N1. Blunted affect; N2. Emotional withdrawal; N3. Poor rapport; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity; G7. Motor retardation; and G16. Active social avoidance).
  Participants are rated from 1 to 7 on each symptom subscale. Higher score indicates more severe symptoms. The negative symptoms in schizophrenia are the diminution or loss of normal functions.
Time Frame: At baseline and week 52
Population: All treated participants with baseline and week 52 PANSS marder factor negative scores.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | KarXT
Number analyzed (Participants) | 558
Score on a Scale | -1.1 (4.49)

8. Secondary Outcome: Change From Baseline in Clinical Global Impressions-severity (CGI-S) Score Week 52
Description: Completed independently by a clinician, the CGI-S categorizes the severity of the illness as: 1 = Normal, not at all ill; 2 = Borderline mentally ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; and 7 = Among the most extremely ill patients, by asking the clinical 1 question and providing a rating based upon observed and reported symptoms, behavior, and function in the past 7 days to reflect the average severity level across the 7 days. Higher score indicates more severe illness.
Time Frame: At baseline and week 52
Population: All treated participants with baseline and week 52 clinical global Impressions-severity (CGI-S) scores.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | KarXT
Number analyzed (Participants) | 283
Score on a Scale | -0.4 (0.70)

9. Secondary Outcome: Percentage of Participants With a ≥30% Reduction in PANSS Total Score at Week 52
Description: A PANSS responder is defined as a participant with a reduction from baseline of at least a 30% improvement at Week 52 in the PANSS total score. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. PANSS total score is the sum of all 30 items with a minimum score of 30 and a maximum score of 210. Higher scores indicate more severe symptoms.
Time Frame: At baseline and week 52
Population: All treated participants with baseline and week 52 PANSS total scores.
Measure: Number; unit: percentage of participants
Arm/Group | KarXT
Number analyzed (Participants) | 283
percentage of participants | 9.2

10. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)
Description: LFT elevations, inclusive of drug-induced liver injury (DILI) and symptomatic orthostasis including syncope (a transient loss of consciousness or fainting) is to be captured as an AESI and reported as such. Non symptomatic orthostasis will not be reported as an AESI. Any such AESI due to any cause, whether or not related to KarXT, must be reported within 24 hours of occurrence or when the investigator becomes aware of the event.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 566
Participants | 19

11. Secondary Outcome: Number of Participants With Anticholinergic and Procholinergic Symptoms
Description: The number of participants experiencing adverse events related to procholinergic symptoms (believed to be associated with xanomeline) and anticholinergic symptoms (believed to be associated with trospium) symptoms. Examples of procholinergic symptoms include vomiting, nausea, diarrhea, sweating and hyper-salivation. Examples of anticholinergic include dizziness, confusion, hallucinations, and somnolence.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 566
Participants
  Anticholinergic | 159
  Procholinergic | 210

12. Secondary Outcome: Change From Baseline in Simpson-Angus Rating Scale (SAS)
Description: The Simpson-Angus Rating Scale (SAS) is a clinical tool used to assess the severity of extrapyramidal symptoms (EPS), which are drug-induced movement disorders often associated with antipsychotic medications. The scale consists of 10 items, each rated from 0 (none) to 4 (severe), with a total score range of 0 to 40.
  Higher scores indicate more severe symptoms.
  The SAS helps clinicians monitor and manage EPS in patients, guiding treatment decisions to minimize these side effects.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: All treated participants with baseline and at least one post-baseline SAS score.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | KarXT
Number analyzed (Participants) | 404
Score on a Scale | 0.1 (0.48)

13. Secondary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS)
Description: The BARS for akathisia is a rating scale used to assess the severity of drug-induced akathisia, or restlessness, involuntary movements and inability to sit still. The range of scores is 0 to 14, with higher scores indicating greater severity.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: All treated participants with baseline and at least one post-baseline BARS score.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | KarXT
Number analyzed (Participants) | 405
Score on a Scale | 0.1 (0.58)

14. Secondary Outcome: Change From Baseline in Total Abnormal Involuntary Movement Scale (AIMS)
Description: The Abnormal Involuntary Movement Scale (AIMS) is a tool used to assess the severity of tardive dyskinesia and other involuntary movements, often caused by antipsychotic medications. It includes 12 items, with the first 10 focusing on specific body areas and movement severity, rated from 0 (none) to 4 (severe).
  The total score ranges from 0 to 28, with higher scores indicating more severe symptoms.
  AIMS helps clinicians monitor and manage these movement disorders, guiding treatment adjustments to reduce side effects.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: All treated participants with baseline and at least one post-baseline AIMS score.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | KarXT
Number analyzed (Participants) | 566
Score on a Scale | 0.1 (0.57)

15. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: BMI is a person's weight in kilograms divided by the square of height in meters. Baseline is defined as measurements taken at screening.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: All treated participants with baseline and at least one post-baseline BMI results.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | KarXT
Number analyzed (Participants) | 408
kg/m^2 | -0.761 (2.0108)

16. Secondary Outcome: Change From Baseline in Waist Circumference
Description: The change in waist circumference in centimeters from baseline. Baseline is defined as measurements taken at screening.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: All treated participants with baseline and at least one post-baseline waist circumference results.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | KarXT
Number analyzed (Participants) | 403
cm | -1.549 (7.3558)

17. Secondary Outcome: Change From Baseline in Blood Pressure Values
Description: The change from baseline in orthostatic diastolic and systolic blood pressure measured while supine and standing after 2 minutes.
  Baseline is defined as measurements taken at screening.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: All treated participants with baseline and at least one post-baseline blood pressure results.
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | KarXT
Number analyzed (Participants) | 408
mmHG
  Supine Systolic | 0.1 (12.83)
  Standing Systolic | -0.7 (12.33)
  Supine Diastolic | 0.1 (8.72)
  Standing Diastolic | -0.2 (8.26)

18. Secondary Outcome: Change From Baseline in Heart Rate
Description: The change from baseline in orthostatic heart rate measured while supine and standing after 2 minutes. Baseline is defined as measurements taken at screening.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: All treated participants with baseline and at least one post-baseline heart rate results.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | KarXT
Number analyzed (Participants) | 408
beats/min
  Supine Heart Rate | 0.7 (11.43)
  Standing Heart Rate | 0.1 (11.22)

19. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Assessments
Description: Laboratory assessments include:
  * Hematology
  * Serum chemistry
  * Urinalysis
  * HbA1c
  * Prolactin levels
  * Coagulation studies
  * Viral Serology
  * Pregnancy test
Time Frame: From time of consent to end of study (approximately 400 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 566
Participants | 0

20. Secondary Outcome: Number of Participants With Clinically Significant Changes in 12 Lead Electrocardiogram
Description: An electrocardiogram (ECG) measures electrical activity of the heart to detect cardiac problems.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 566
Participants | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination
Description: A complete physical examination (body temperature, general appearance, head/eyes/ears/nose/throat [HEENT], examination of thorax and abdomen, assessment of cardiac, musculoskeletal, and circulatory systems, palpations for lymphadenopathy, and limited neurological examination) will be performed.
  A targeted physical examination includes at a minimum body temperature, a check of general appearance, as well as examination of organ systems that are relevant to the investigator based on review of the participant's reported AEs, review of systems, or concomitant medication use. These also include symptom-driven physical examinations which will be performed as clinically indicated at any study visit.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 566
Participants | 3

22. Secondary Outcome: Number of Participants With Suicidal Ideation Based on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) is a tool used to assess the severity and immediacy of suicidal ideation and behavior. It covers suicidal thoughts, plans, and actions, including the frequency, intensity, and context of these behaviors. The C-SSRS does not use a numerical scoring system like some other assessment tools. Instead, it categorizes the severity of suicidal ideation and behavior based on specific criteria. The scale helps clinicians identify individuals at risk of suicide and monitor changes over time, guiding treatment decisions and ensuring safety. It is quick and easy to administer, making it useful in various clinical and research settings.
Time Frame: From time of consent to end of study (approximately 400 days)
Population: All treated participants with C-SSRS results.
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 406
Participants
  Wish to be dead | 1
  Non-Specific Active Suicidal Thoughts | 1
  Active Suicidal Ideation with any methods without intent to act | 0
  Active Suicidal Ideation with some intent to act but without a plan | 1
  Active Suicidal Ideation with specific plan and intent | 0

ADVERSE EVENTS:
Time Frame: From time of consent to end of study (approximately 400 days)
Description: The number at Risk for All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | KarXT
All-Cause Mortality (participants affected / at risk) | 2/566
Serious Adverse Events (participants affected / at risk) | 41/566
Other Adverse Events (participants affected / at risk) | 356/566
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KarXT (N=566)
Angina pectoris (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Death (General disorders) | 2
COVID-19 (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Burns third degree (Injury, poisoning and procedural complications) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Depressive symptom (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 4
Schizophrenia (Psychiatric disorders) | 10
Suicide attempt (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Psychosocial support (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KarXT (N=566)
Constipation (Gastrointestinal disorders) | 102
Diarrhoea (Gastrointestinal disorders) | 52
Dry mouth (Gastrointestinal disorders) | 53
Dyspepsia (Gastrointestinal disorders) | 41
Nausea (Gastrointestinal disorders) | 131
Vomiting (Gastrointestinal disorders) | 113
Weight decreased (Investigations) | 32
Dizziness (Nervous system disorders) | 49
Headache (Nervous system disorders) | 46
Somnolence (Nervous system disorders) | 35
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 29
Hypertension (Vascular disorders) | 59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT04820309/Prot_SAP_000.pdf